CLINICAL TRIAL: NCT06742333
Title: Early Intervention in Plaque Psoriasis: is Bimekizumab Able to Delay Chronic Inflammation? Prospective Multicenter Interventional Study
Brief Title: Early Intervention in Plaque Psoriasis: is Bimekizumab Able to Delay Chronic Inflammation?
Acronym: EARLYPSO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-PP-01
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — bimekizumab; Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group Bimekizumab (Experimental): Bimekizumab 320mg given at weeks wk0, wk4, wk8 and wk12
  Interventions: Drug: Bimekizumab
- Comparator group Clobetasol (Active Comparator): Once daily evening application of 0.05% of clobetasol ointment for up to 4 weeks. The randomization will take place at the end of V1, baseline visit, after verifying the selection criteria and written consent, by the investigator in charge of the patient in each center.
  Interventions: Drug: Clobetasol

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab 320mg given at weeks wk0, wk4, wk8 and wk12
  Arms: Treatment Group Bimekizumab
Drug: Clobetasol — Once daily evening application of 0.05% of clobetasol ointment for up to 4 weeks
  Arms: Comparator group Clobetasol

SUMMARY:
Psoriasis is a chronic inflammatory condition driven by a complex interplay between heritable and microenvironmental factors. Genome-wide heritability for psoriasis (PsO) is estimated at up to 50%. Although bearing genetic susceptibility at birth, most patients will remain disease free for years until an exposomal trigger activates the immunological pathway that leads to the first disease flare. In rare patients, the first flare is an isolated event, but in most patients it will evolve into a chronically relapsing-remitting disease characterized by lasting lesions and recurrent flares. Primary objective is to compare efficacy of bimekizumab versus topical corticosteroids on psoriasis clinical disease activity, assessed by PGA, at week 16 and week 24.

Patients will be randomized 1:1 to receive either 320mg bimekizumab at weeks 0 (W0), W4, W8 and W12, or clobetasol ointment for 2 to 4 weeks until complete clearance of the lesion. After a maximum of 4 weeks topical clobetasol will be applied twice weekly on the site of lesion until week 16 then stopped. Patients will not receive active treatment between week 16-24. Between week 24-96 patients that flare can receive continuous topical clobetasol if needed. These patients will be considered non-responders at subsequent timepoints for the main analysis. If the patients worsen their psoriasis under the treatments given during the study and progress to moderate or severe psoriasis (PASI 10 and above) they will end their participation to the study to receive a treatment adapted to the new severity of their psoriasis. The patients will be referred to their dermatologist to receive the actual standard of care adapted to their new condition.

During the study, the following assessments will be performed and samples will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. ≥ 18 and <45 years
3. Plaque psoriasis without psoriatic arthritis
4. Patients with mild psoriasis PASI >2 and <6
5. Patient with at least one lesion on the elbows, or the knees, or the lower back to be recorded as target lesion (additional lesions in other areas on top are allowed)
6. Disease duration less than 6 months (short duration psoriasis) or >2 years (long duration psoriasis)
7. The psoriasis lesions should not having being treated by any topical treatment for at least 2 weeks
8. For women of childbearing potential, an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study. A urine pregnancy test (βHCG in urines) will be performed.

   Thus, a woman who is permanently sterile and therefore unable to procreate should not be subjected to pregnancy tests.

   Women who are sexually abstinent are not requested to use a contraception. However, they must agree to take one if they want to become sexually active.
9. Affiliation to a social security system
10. Signed informed consent
11. Patient willing and able to attend all study visits

Exclusion Criteria:

1. Pregnant or breast-feeding women. Or women who plan to get pregnant during the study duration.
2. Concomitant use of topical or systemic immunosuppressive medication or steroids in the past 12 weeks
3. Personal history of skin cancer
4. Personal history of cancer of less than 5 years
5. Patients with active infection
6. Abnormal blood counts (neutrophils <1500/mm3 and platelets <150 000/mm3) and/or positive HIV, HVB and HVC testing at screening.
7. Patients with personal history of keloid scars
8. Patients with personal history of hypersentitivity to xylocaine and/or adrenalin
9. Vulnerable people: minors, adult under guardianship or deprived of freedom
10. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2028-07-22 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of bimekizumab versus topical corticosteroids on psoriasis | at 24 weeks
  The Physician's global Assessment is a validated method to simply assess plaque psoriasis severity using a scale ranging from 0 to 5 (Low to severe)

SECONDARY OUTCOMES:
To compare patient's quality of life between BKZ and topical corticosteroids | at 24 weeks
  The Dermatological Life Quality Index is the main score to assess the impact of dermatoses on the quality of life of affected individuals. The score ranges from 0 to 30, with quality of life varying from pleasant to not at all pleasant.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Passeron, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (7):
- France (7):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Saint-Joseph, Marseille
  - Cabinet Dermatologie Dr RUER, Martigues
  - CHU Saint-Etienne, Saint-Etienne
  - CHITS, Toulon
  - Médipole Villeurbanne, Villeurbanne

IPD SHARING:
Plan to Share IPD: No